CLINICAL TRIAL: NCT01382017
Title: Effects of Lacosamide on Human Motor Cortex Excitability: a Transcranial Magnetic Stimulation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Nicolas Lang, PD Dr. med., University of Kiel
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LCM-TMS-2010
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Healthy Male Volunteers
Keywords: lacosamide; carbamazepine; placebo; transcranial magnetic stimulation; TMS; motor cortex; sodium channel; inhibition; threshold
MeSH Terms: conditions — Inhibition, Psychological | interventions — Lacosamide; Carbamazepine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo
- Lasosamide 200 (Experimental): Lacosamide 200 mg
  Interventions: Drug: Lacosamide
- Lacosamide 400 (Experimental): Lacosamide 400 mg
  Interventions: Drug: Lacosamide
- Carbamazepine 600 (Active Comparator): Carbamazepine 600 mg
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Lacosamide — Lacosamide 200 or 400 mg
  Arms: Lacosamide 400; Lasosamide 200
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Carbamazepine — Carbamazepine 600 mg
  Arms: Carbamazepine 600

SUMMARY:
This study has been designed to explore dose-depended effects of lacosamide (LCM) on motor cortex excitability with TMS in a randomized, double-blind, placebo-controlled crossover trial in young healthy human subjects, and to compare the pattern of excitability changes induced by LCM with those of carbamazepine (CBZ). LCM selectively enhances slow inactivation of voltage-gated sodium channel, and, in contrast to CBZ, does not affect steady-state fast inactivation (Errington et al., 2006). The enhancement of slow inactivation of sodium channels by LCM is a novel manner to modulate sodium channels and leads to normalization of activation thresholds and a reduced pathophysiological hyper-responsiveness, thereby effectively controlling neuronal hyperexcitability without affecting physiological activity (Beyreuther et al., 2007). Therefore, it is thought that LCM, compared to CBZ, will be better tolerated in clinical settings while being as or even more effective in controlling seizure activity. On the basis of the results from nonhuman studies, it is hypothesized that the TMS profile of LCM will be distinguishable from that of CBZ. CBZ, like other 'classical' sodium channel blockers such as phenytoin, predominantly demonstrated elevated TMS motor thresholds indicating reduced neuronal membrane excitability, without developing significant changes of synaptic intracortical inhibition and facilitation (Ziemann et al., 1996; Chen et al., 1997; Lee et al., 2005). Because of its novel mode of action it can only be speculated which TMS parameters LCM might affect. For example, more than exclusively affecting neuronal membrane excitability, LCM could possibly also affect inhibitory mechanisms such as short- and long-latency intracortical inhibition (Valls-Sole et al., 1992; Kujirai et al., 1993). This would in line with other well-tolerated modern antiepileptic drugs (Ziemann et al., 1996; Reis et al., 2002; Lang et al., 2006).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* male
* right-handed
* aged 18-45 years

Exclusion Criteria:

* cardiac pacemaker
* metal implants in the head
* intake of any medication
* previous neurologic, psychiatric, or chronic internal diseases
* pregnancy or breastfeeding; drug, nicotine, or alcohol abuse
* known or expected intolerance to soy beans, peanuts, LCM or CBZ; abnormal ECG with prolonged PQ-interval
* participation in another clinical trial within the previous 8 weeks

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
TMS measures of cortical excitability | within 24h after intake of study medication
  Transcranial magnetic stimulation (TMS) measurements included resting motor thresholds (RMT) and active motor thresholds (AMT), the intensity to evoke MEP of ∼1mV peak-to-peak amplitude (SI1mV), short-interval intracortical inhibition/intracortical facilitation (SICI/ICF), long-interval intracortical inhibition (LICI), short-interval intracortical facilitation (SICF), recruitment curves, MEP under tonic activation (aMEP), and cortical silent period (CSP), and MEP changes in response to short trains of repetitive TMS.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Lang, PD Dr. med., Principal Investigator — Christian-Albrechts University Kiel, Germany
Locations (1):
- Departmenr of Neurology, UKSH Campus Kiel, Kiel, Germany

REFERENCES:
- See also: Department of Neurology, University of Kiel, Germany — http://www.uksh.de/neurologie-kiel